CLINICAL TRIAL: NCT00681772
Title: Open-label, Multi-centre, Study to Investigate the Safety, Tolerability and Efficacy of Flexible Doses of Vardenafil Given on Demand in Males With Erectile Dysfunction
Brief Title: Evaluation of the Safety and Efficacy of Vardenafil in Subjects With Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Healthcare AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100541
Record Dates: First submitted 2008-04-18; First posted 2008-05-21 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 5mg, 10mg or 20mg taken 1 hours before sexual intercourse

SUMMARY:
Erectile dysfunction (ED) is defined as the inability to achieve or maintain an erection sufficient for satisfactory sexual performance. An ideal treatment option should be effective and reliable, have minimal side effects, be simple to use and affordable. The aim of this study was to investigate safety, tolerability and efficacy of vardenafil following a flexible dose treatment schedule in subjects with varying aetiology.

ELIGIBILITY:
Inclusion Criteria:

* Men >/= 18 years of age,
* ED 6 months or longer
* Stable sexual relationship for > 6 month.

Exclusion Criteria:

* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within prior 6 month
* Nitrate therapy
* Other exclusion criteria apply according to the Summary of Product Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2003-03; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function - Erectile Function Domain | 12 weeks

SECONDARY OUTCOMES:
Sexual Encounter Profile Question 2 and 3 | 12 weeks
Global Assessment Question | 12 weeks
Other diary based variables | 12 weeks
Safety and tolerability | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer